CLINICAL TRIAL: NCT00809029
Title: The Influence Of GIP (Glucose-Dependent Insulinotropic Polypeptide) Infusion On Hormone Sensitive Lipase, Lipoprotein Lipase And Adipokine Expression In Human Subcutaneous Adipose Tissue: An In Vivo Study
Brief Title: The Influence Of GIP (Glucose-Dependent Insulinotropic Polypeptide) Infusion On Human Adipose Tissue: An In Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, DR CHRISTINA DAOUSI, Clinical Senior Lecturer, Liverpool University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 08/H1001/20; 08DE001
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Adipose Tissue
Keywords: GIP; OBESITY; HSL; LPL; ADIPOCYTOKINES; BARIATRIC SURGERY
MeSH Terms: conditions — Obesity | interventions — Gastric Inhibitory Polypeptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: GIP (glucose dependent insulinotropic peptide) infusion — an intravenous infusion of GIP (glucose dependent insulinotropic peptide)or placebo will be administered at a rate of 2 pmol/kg/min and maintained for 240 minutes.
  Other Names: GIP (glucose dependent insulinotropic peptide)

SUMMARY:
Study part-1

GIP (glucose-dependent insulinotropic polypeptide) is one of the two main incretin hormones secreted by specialized cells of the gastrointestinal tract in response to ingestion of nutrients. Data emerging from studies in animal models and cultured human fat cells support a physiological role for GIP in the adipose tissue metabolism which may contribute to the pathogenesis of obesity.

The proposed study will shed more light on the interactions between gut hormones and adipose tissue. For this pilot study, male subjects fulfilling the inclusion criteria will be given GIP or placebo infusions in a randomized manner. Fat tissue biopsies will be obtained from all subjects during both visits, once in the basal state (before the start of the peptide/placebo infusion) and then repeated at the end of the period of infusion.

Study part-2

Surgery represents the most effective therapeutic modality for morbid obesity. Resolution of type 2 diabetes mellitus (T2DM) has been consistently observed as an additional benefit of surgical treatment of obesity. The mechanisms underlying the dramatic effects of surgery on insulin sensitivity and β-cell function are poorly understood. Bariatric surgery (gastric bypass) promotes changes in the enteroendocrine system as a result of nutrient diversion from the physiological intestinal routes with subsequent profound modification of gut hormone secretion

We hypothesize that restoration of GIP action after bariatric procedures plays a cardinal role in the improvement and/or restoration of diabetes, we propose to study patients (both sex)with morbid obesity and T2DM within 3 months after their surgery. Their responses will be compared to those of BMI matched control subjects with normal glucose tolerance

ELIGIBILITY:
Inclusion Criteria:

* Lean (BMI 20-25 kg/m2) subjects with normal glucose tolerance
* Obese (BMI >30 kg/m2) subjects also with normal glucose tolerance.
* Obese with impaired glucose tolerance
* Obese with diet controlled diabetes mellitus
* Morbid obesity, type diabetes and post bariatric surgery (study part 2)

Exclusion Criteria:

* History of severe cardiac, hepatic or renal disease
* Thyroid dysfunction (hyper-or hypothyroidism), or other endocrine disturbance (acromegaly, growth hormone deficiency, hypoadrenalism or cortisol overproduction)
* Current malignant disease
* Known alcohol misuse
* Major psychiatric disease (including current use of antidepressants)
* History of major eating disorder (anorexia or bulimia nervosa)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To measure Lipoprotein lipase (LPL) and Hormone sensitive Lipase (HSL) activity in adipose tissue | Before and after 4 hours of infusion

SECONDARY OUTCOMES:
To determine the role of GIP in adipocytokine gene expression and secretion from human subcutaneous adipose tissue | Baseline and after 4 hours of continuous infusion

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTINA DAOUSI, MD FRCP, Principal Investigator — UNIVERSITY HOSPITAL AINTREE NHS TRUST
Locations (1):
- University Hospital Aintree, Liverpool, United Kingdom